CLINICAL TRIAL: NCT03643783
Title: Impact of Plasma Soluble Prorenin Receptor in Obese and Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Tulane University Health Sciences Center (Other); UAB-CCTS Network Mulitdisciplinary Pilot Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-374
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Type2 Diabetes; Bariatric Surgery Candidate
Keywords: Bariatric Surgery; Prorenin; Hypertension; Obesity
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric Obese Patients: Obese patients, including men and women, White (Caucasians), Africa American, and Hispanic or Latino racial categories, and ages 18-70 years, who are enrolled and planning to undertake bariatric surgery in the Outpatient Bariatric Surgery Clinic at Tulane University, HSC (Christopher G. Ducoin, MD, MPH; Chair of Bariatric Surgery Clinic and Surgeon, and Shauna Levy, MD, Bariatric Surgeon Specialist).
- Lean Control Patients: Plasma samples from lean control patients that have already been collected and are available as part of the Tulane Obesity-Endocannabinoids Study (Tina Thethi, M.D, Collaborator).

SUMMARY:
Obesity increases the risk for type 2 diabetes mellitus, high blood pressure, and mortality. Obesity is a major health problem in the United States, especially in the Deep South regions. Obesity increases the risk for T2DM, the occurrence of hypertension, and mortality; but the efficacy of long-term weight loss medications has been disappointing. There are three options available for patients who want to lose weight: lifestyle modification, pills, or weight loss by bariatric surgery. When we compare the three options available, bariatric surgery is the most effective method to lose weight at present. Bariatric surgery allows patients lose the most weight, be able to sustain the weight reduction over time and, more importantly, diabetes mellitus and other cardiovascular risk factors significantly improve. Understanding the link among obesitydiabetes-hypertension is crucial in order to develop new therapeutic targets to decrease CVD morbidity and mortality. There is less prevalence of coronary artery disease (CAD) in premenopausal women than in men, but, once initiated, the morbidity and mortality due to CAD in women is worse than in men, thus highlighting this sex difference in CVD. Indeed, women with diabetes exhibit a higher risk of myocardial infarction and stroke mortality than men, compared to people without diabetes. In obese subjects, there is inappropriate activation of the systemic and adipose renin-angiotensin system. The prorenin receptor is a molecule expressed in various tissues including fat tissue and part of it, the soluble prorenin receptor, can be secreted into the blood. The prorenin receptor is part of a very important system that regulates blood pressure and fat in our body, the renin-angiotensin system. In this prospective observational human pilot study, we will determine whether the adipose tissue is the major supplier of soluble prorenin receptor levels in the plasma of obese patients and the relationship between blood soluble prorenin receptor and diabetes mellitus, obesity, high blood pressure and other important cardiovascular risk factors. Outcomes from this study will allow a better understanding of the complex factors that link obesity, diabetes mellitus, and other cardiovascular risk factors and designing better therapeutic alternatives to improve patient's health, particularly in obese diabetic women.

DETAILED DESCRIPTION:
Human blood samples will be collected prospectively from 50 obese patients, who are enrolled and planning to undertake bariatric surgery in the Outpatient Bariatric Surgery Clinic at Tulane University, HSC (Christopher G. Ducoin, MD, MPH; Chair of Bariatric Surgery Clinic and Surgeon, and Shauna Levy, MD, Bariatric Surgeon Specialist). Type of bariatric surgery used in each patient will be recorded. Because it has been shown that after 6 months of bariatric surgery, there is about 50-60% BW loss 15-18, we plan to obtain two tubes of blood samples with 5 mL of blood each. Blood will be drawn during the pre-Op visit and during 3 visits following the bariatric surgery: 1 week ± 2-3 days, 1 month ± 2 weeks and 6 months ± 1 - 2 months. Blood samples will be used for plasma measurements of: glycaemia, HbA1c, lipids profile (LDL, HDL,triglycerides) and sPRR. Time of drawing of blood sample will be recorded due to potential effects of circadian rhythms to the RAS. Quantification of plasma sPRR by ELISA will be performed in Dr. Minolfa Prieto's laboratory located at Tulane University School of Medicine. Patient biological samples will be identified by a code that will link the sample to the patient. After conclusion of the study, samples will be used exclusively for obesity and T2DM related conditions research. Background Factors will include: sex, age, race, ethnicity, health insurance status, and personal medical history will assess presence of any of the following conditions: diabetes mellitus or hypertension (including any of the following treatments: antihypertensive drugs -ACEi, AT1R blockers, diuretics, or calcium antagonists), use of oral contraceptives or hormone replacement, previous surgeries (type, date), last menstruation date including any menstrual irregularity, congestive heart failure (CHF), peripheral vascular disease (PVD), pulmonary hypertension (PHTN), or ischemic heart disease, obstructive sleep apnea (OSA), asthma, deep vein thrombosis/pulmonary embolism (DVT/PE), gastroesophageal reflux disease (GERD), liver disease, dyslipidemia, polycystic ovarian syndrome, depression, alcohol use, substance abuse, and/or tobacco use. Physical exam will include: BW, BMI, waist circumference, height, office BP (DBP and SBP measured at the Outpatient Clinic with the patient in a sitting position after resting for at least 5 min), and pulse rate Patient biological samples will be identified by a code linking the sample with the patient. Plasma samples for ELISA measurements will be assayed in duplicate in a blinded fashion. ELISA kits are commercial available and manufactured by IBL America, Inc. This assay is routinely performed in the PI's laboratory and has been validated using appropriate standards (provided by the manufacturers). We will use duplicate or triplicate samples when assayed. Biological controls such as buffer as blank will be used as technical controls. Because ELISA kits will be obtained from commercial vendors, authentication by the vendor(s) includes certifications of reactivity, purity, applications. These methods and outcomes have been previously reported. Internal controls standards curve of various concentrations of sPRR will be included in each plate reading for comparison purposes. To reduce bias, samples will be randomly assayed wherever possible and include positive standard controls with known concentrations for comparisons purposes. Both, a data handling plan (outliers, report of missing data) and a statistical analysis plan (Statistical analysis plan, endpoints [primary and secondary], inclusion for multiple testing will be used.. Our lab has authenticated sPRR ELISA and compared with measurements published by others. To ensure the detection of meaningful and realistic differences, the sample numbers are based on the requirement to perform each assay (Power and Sample size calculations). To ensure reproducibility, all protocols will be reported including all of the experimental conditions in detail. After conclusion of the study, samples will be used exclusively for obesity and DM related research. Aim 1: Determine whether plasma levels of sPRR decrease in obese patients after bariatric surgery. Scientific Premise and Rationale: In obese rats, PRR and renin are augmented two-fold in adipose tissue. Preliminary data from mice with T2DM-induced by high fat diet showed presence of a phenotype characterized by obesity, increased SBP, glucose intolerance, marked insulin resistance, and increased levels of sPRR in plasma by 18-wks on the dietary regimen. These mice also showed increased PRR expression in adipocytes from visceral fat. Our preliminary study showed that plasma sPRR levels are higher in lean men than lean women. In contrast, plasma sPRR levels were higher in obese diabetic women than in men. Furthermore, we found that obese patients with T2DM exhibited a positive correlation between plasma sPRR and BMI in women but not in men. This aims seeks to test the hypothesis that adipose tissue is the major supplier of plasma sPRR in obese patients.

Experimental Design: quantifications will be done in plasma samples obtained from 50 obese patients undergoing bariatric surgery. Plasma samples will be drawn before bariatric surgery (pre-Op visit) and at each of 2 follow-up visits (1 month ± 1 - 2 weeks and at 6 months ± 1-2 months) for the assessment of plasma sPRR by ELISA (Prieto's Lab, Tulane University) (See Power Analysis). These samples will be obtained from patients of the Bariatric and Minimal Invasive Surgery Clinic of Christopher G. Ducoin, MD at Tulane HSC (Collaborator). Comparisons will be established with human biological de-identified plasma samples from lean control patients that have already been collected and are available as part of the Tulane Obesity-Endocannabinoids Study (Tina Thethi, M.D, Collaborator). After patient's consent agreement, the patient will be examined in the Bariatric and Minimal Invasive Surgery Clinic for vital signs, BP (SBP and DBP, taken by sphygmomanometry), waist-to-hip ratio, and BMI. Fasting blood samples will be drawn by vein puncture for glycaemia, HbA1c, lipids profile (LDL, HDL, triglycerides), and sPRR. Background factors and personal medical history will be taken as described in the Study Design section. Power Analysis and Statistical Considerations: All the outcomes at each time point will be summarized as mean and standard deviation (SD). The repeated measures analysis of variance and paired test will be conducted to evaluate the change across the time points. The historical data suggest that about 10 patients receive bariatric surgery per month in the Outpatient Bariatric Clinic at Tulane University; we expect that at least 50 eligible patients will be recruited in the first 6 months of this project.

Aim 2: Define whether changes in plasma levels of sPRR correlate with improvement of T2DM parameters in obese patients subsequent to weight loss after bariatric surgery. Scientific Premise and Rationale: Obesity and T2DM are major risk factors for CVD.

Activation of RAS is implicated in the pathogenesis of CV risk factors. Often T2DM is improved immediately after bariatric surgery and even further with the sustained substantial BW loss. However, it remains unknown whether adipose tissue is the major supplier of sPRR in the plasma of obese patients, and if plasma sPRR contributes to T2DM and CV complications in these patients. Use of sPRR inhibitors would constitute a novel therapeutic approach to manage obesity in women and CV complications. We will test the hypothesis that decreases in levels of plasma sPRR after bariatric surgery is associated with the improvement in glycemic control and lipid profile in obese patients. Analysis and Statistical Considerations: Multiple linear regression models will be used to measure the association between sPRR, glycaemia, HbA1c, lipids profile (LDL, HDL, triglycerides). Comparisons will be established with values before and 2 visits after surgery. The proposed n=50 will be sufficient to fit models with up to 7 predictors and to have 80% power to detect a significant association between sPRR and any one predictor if at least 12.25% of the total variability of sPRR is accounted for by the predictor. Unadjusted and adjusted correlations and associated P values will be reported.

Expected Results, Pitfalls, and Alternative Approach Aim 1: To our knowledge, no previous study has defined the relationship among plasma sPRR-obesity-T2DM or has established the correlations between plasma sPRR and BMI, WHR, or HbA1c. We expect that plasma sPRR levels will be higher in obese than in lean control samples, and that compared with control, plasma sPRR levels will be higher in T2DM obese patients. We anticipate that plasma sPRR levels will be positively associated with obesity in T2DM obese women but not in male counterparts after adjusting for background factors, suggesting that increases in plasma sPRR in women might be due to hyperandrogenemia. Aim 2: will define whether changes in plasma sPRR correlate with the improvement of T2DM and lipid profile in obese patients after bariatric surgery. Based on our strong preliminary data, we anticipate that the outcomes will allow better understanding of the role of sPRR and metabolic risk factors in obese patients. Potential pitfalls: Because patients undergoing bariatric surgery are more commonly women, if recruitment/enrollment of men results to be low, we will justify the analysis with women to men frequency data ratio of 4:1.19 Alternative Approach: We expected that the outcomes allow comparing the impact of the direct effects of the bariatric surgery vs. the long-term effects (probably related to weight loss) on plasma sPRR and insulin resistance. If recruitment is less than expected, we will reach out to other local bariatric surgery centers,including Ochsner Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-70 years of age
* Scheduled to undergo bariatric surgery
* Obese (defined as BMI >=30)

Exclusion Criteria:

* History of hemorrhagic stroke or myocardium infarction in the previous 6 months.
* Women who are currently pregnant
* Diagnosed with a malignant disease
* Uncontrolled diabetes mellitus (defined as HbA1c>10.0%)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese men and women of all races between the ages of 18-70 who are scheduled to undergo bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels of sPRR | 1 month and 6 months postop
  Determine whether changes in plasma levels of sPRR decrease in obese patients after bariatric surgery.
Change in T2DM parameters and sPRR after surgery | 1 month and 6 months postop
  Define whether changes in plasma levels of sPRR correlate with improvement of T2DM parameters in obese patients subsequent to weight loss after bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Minolfa Prieto, MD PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Fryar CD, Flegal KM. Prevalence of Obesity Among Adults and Youth: United States, 2011-2014. NCHS Data Brief. 2015 Nov;(219):1-8. PMID 26633046
- [Background] Stamataki KE, Spina J, Rangou DB, Chlouverakis CS, Piaditis GP. Ovarian function in women with non-insulin dependent diabetes mellitus. Clin Endocrinol (Oxf). 1996 Nov;45(5):615-21. doi: 10.1046/j.1365-2265.1996.00795.x. PMID 8977760
- [Background] Engeli S, Schling P, Gorzelniak K, Boschmann M, Janke J, Ailhaud G, Teboul M, Massiera F, Sharma AM. The adipose-tissue renin-angiotensin-aldosterone system: role in the metabolic syndrome? Int J Biochem Cell Biol. 2003 Jun;35(6):807-25. doi: 10.1016/s1357-2725(02)00311-4. PMID 12676168
- [Background] Nguyen G, Delarue F, Berrou J, Rondeau E, Sraer JD. Specific receptor binding of renin on human mesangial cells in culture increases plasminogen activator inhibitor-1 antigen. Kidney Int. 1996 Dec;50(6):1897-903. doi: 10.1038/ki.1996.511. PMID 8943472
- [Background] Cousin C, Bracquart D, Contrepas A, Corvol P, Muller L, Nguyen G. Soluble form of the (pro)renin receptor generated by intracellular cleavage by furin is secreted in plasma. Hypertension. 2009 Jun;53(6):1077-82. doi: 10.1161/HYPERTENSIONAHA.108.127258. Epub 2009 Apr 20. PMID 19380613
- [Background] Nguyen G, Muller DN. The biology of the (pro)renin receptor. J Am Soc Nephrol. 2010 Jan;21(1):18-23. doi: 10.1681/ASN.2009030300. Epub 2009 Nov 16. PMID 19917780
- [Background] Achard V, Tassistro V, Boullu-Ciocca S, Grino M. Expression and nutritional regulation of the (pro)renin receptor in rat visceral adipose tissue. J Endocrinol Invest. 2011 Dec;34(11):840-6. doi: 10.3275/7627. Epub 2011 Apr 6. PMID 21483231
- [Background] Wu CH, Mohammadmoradi S, Thompson J, Su W, Gong M, Nguyen G, Yiannikouris F. Adipocyte (Pro)Renin-Receptor Deficiency Induces Lipodystrophy, Liver Steatosis and Increases Blood Pressure in Male Mice. Hypertension. 2016 Jul;68(1):213-9. doi: 10.1161/HYPERTENSIONAHA.115.06954. Epub 2016 May 16. PMID 27185751
- [Background] Hu E, Kim JB, Sarraf P, Spiegelman BM. Inhibition of adipogenesis through MAP kinase-mediated phosphorylation of PPARgamma. Science. 1996 Dec 20;274(5295):2100-3. doi: 10.1126/science.274.5295.2100. PMID 8953045
- [Background] Morimoto S, Ando T, Niiyama M, Seki Y, Yoshida N, Watanabe D, Kawakami-Mori F, Kobori H, Nishiyama A, Ichihara A. Serum soluble (pro)renin receptor levels in patients with essential hypertension. Hypertens Res. 2014 Jul;37(7):642-8. doi: 10.1038/hr.2014.46. Epub 2014 Mar 20. PMID 24646643
- [Background] Watanabe N, Bokuda K, Fujiwara T, Suzuki T, Mito A, Morimoto S, Jwa SC, Egawa M, Arai Y, Suzuki F, Sago H, Ichihara A. Soluble (pro)renin receptor and blood pressure during pregnancy: a prospective cohort study. Hypertension. 2012 Nov;60(5):1250-6. doi: 10.1161/HYPERTENSIONAHA.112.197418. Epub 2012 Oct 8. PMID 23045457
- [Background] Deinum J, Ronn B, Mathiesen E, Derkx FH, Hop WC, Schalekamp MA. Increase in serum prorenin precedes onset of microalbuminuria in patients with insulin-dependent diabetes mellitus. Diabetologia. 1999 Aug;42(8):1006-10. doi: 10.1007/s001250051260. PMID 10491762
- [Background] Deinum J, Tarnow L, van Gool JM, de Bruin RA, Derkx FH, Schalekamp MA, Parving HH. Plasma renin and prorenin and renin gene variation in patients with insulin-dependent diabetes mellitus and nephropathy. Nephrol Dial Transplant. 1999 Aug;14(8):1904-11. doi: 10.1093/ndt/14.8.1904. PMID 10462269
- [Background] Ferrara A, Mangione CM, Kim C, Marrero DG, Curb D, Stevens M, Selby JV; Translating Research Into Action for Diabetes Study Group. Sex disparities in control and treatment of modifiable cardiovascular disease risk factors among patients with diabetes: Translating Research Into Action for Diabetes (TRIAD) Study. Diabetes Care. 2008 Jan;31(1):69-74. doi: 10.2337/dc07-1244. Epub 2007 Oct 12. PMID 17934157
- [Background] Sharples AJ, Mahawar K, Cheruvu CVN. Systematic review and retrospective validation of prediction models for weight loss after bariatric surgery. Surg Obes Relat Dis. 2017 Nov;13(11):1914-1920. doi: 10.1016/j.soard.2017.08.009. Epub 2017 Aug 12. PMID 28935199
- [Background] Khorgami Z, Shoar S, Andalib A, Aminian A, Brethauer SA, Schauer PR. Trends in utilization of bariatric surgery, 2010-2014: sleeve gastrectomy dominates. Surg Obes Relat Dis. 2017 May;13(5):774-778. doi: 10.1016/j.soard.2017.01.031. Epub 2017 Jan 25. PMID 28256393
- [Background] Wentworth JM, Cheng C, Laurie C, Skinner S, Burton PR, Brown WA, O'Brien PE. Diabetes Outcomes More than a Decade Following Sustained Weight Loss After Laparoscopic Adjustable Gastric Band Surgery. Obes Surg. 2018 Apr;28(4):982-989. doi: 10.1007/s11695-017-2944-7. PMID 28975466
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy for diabetes--3-year outcomes. N Engl J Med. 2014 May 22;370(21):2002-13. doi: 10.1056/NEJMoa1401329. Epub 2014 Mar 31. PMID 24679060
- [Background] Schwartz J, Bashian C, Kushnir L, Nituica C, Slotman GJ. Variation in Clinical Characteristics of Women versus Men Preoperative for Laparoscopic Roux-en-Y Gastric Bypass: Analysis of 83,059 Patients. Am Surg. 2017 Sep 1;83(9):947-951. PMID 28958273